CLINICAL TRIAL: NCT01405482
Title: Botulin Toxin Type A Injections for Thoracic Outlet Syndrome: A Double-Blind, Randomized Control Trial
Brief Title: Botulinum Toxin Injections for Thoracic Outlet Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Merz Pharmaceuticals (Industry)
Responsible Party: Dr. Heather Finlayson, University of British Columbia - Vancouver Coastal Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H11-00407
Record Dates: First submitted 2011-06-23; First posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Botulinum Toxin Type A; Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum Toxin Type A injection (Active Comparator): Double-blind, randomized, placebo-controlled trial evaluating changes in pain, paresthesias, and function in subjects with TOS before, at six weeks, and four months following injection of BTX-A into the scalene muscles and pectoralis minor muscle under EMG guidance.
  Interventions: Drug: Botulinum Toxin Type A
- Normal Saline (Placebo Comparator): Double-blind, randomized, placebo-controlled trial evaluating changes in pain, paresthesias, and function in subjects with TOS before, at six weeks, and four months following injection of placebo into the scalene muscles under EMG guidance.
  Interventions: Other: Normal Saline injection

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Botulinum Toxin Type A 100 units injected under EMG guidance one time into the anterior,middle scalenes and pectoralis minor muscle
  Other Names: Xeomin
  Arms: Botulinum Toxin Type A injection
Other: Normal Saline injection — 10 cc of Normal Saline will be injected under EMG guidance into the Anterior and Middle Scalenes and Pectoralis Minor muscle of individual diagnosed with Thoracic Outlet Syndrome.
  Other Names: Saline
  Arms: Normal Saline

SUMMARY:
Botulinum toxin type A injected into the anterior and middle scalene muscles will reduce the irritation on the neurovascular structures at the interscalene triangle in subjects with TOS. This will lead to reductions in pain and paresthesias, and improvements in function when compared with injection of placebo.

DETAILED DESCRIPTION:
To assess the effect of Botulinum Toxin Type A (BTX-A) injections into the scalene muscles on pain, paresthesias and function in subjects with TOS.

Hypothesis:

BTX-A injected into the anterior and middle scalene muscles will reduce the irritation on the neurovascular structures at the interscalene triangle in subjects with TOS. This will lead to reductions in pain and paresthesias, and improvements in function when compared with injection of placebo.

Study design:

Double-blind, randomized, placebo-controlled parallel groups effectiveness trial evaluating changes in pain, paresthesias and function before, at six weeks and four months following injection.

Study population:

Sixty subjects at least eighteen years of age with a clinical diagnosis of TOS of at least three months duration but less than one year, referred to our practice for management of TOS.

Intervention:

Each subject will receive an injection under EMG guidance into the anterior and middle scalene muscles of either 100 units of BTX-A (experimental group), or normal saline (control group). Outcome measures:

The primary outcome measure will be pain as measured on a ten point Numeric Rating Scale with a two point reduction considered significant. Secondary outcomes will be paresthesias as measured on a Numeric Rating Scale, function measured on the Disabilities of the arm, shoulder and hand (DASH) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 19 years
* Medically stable
* Able to give informed consent
* Meets criteria for clinical diagnosis of TOS
* Symptoms of TOS present for at least three months and less than two year
* Have had EMG studies and a CT or MRI scan of the cervical spine

Exclusion Criteria:

* Prior treatment with BTX-A
* Allergy to BTX-A
* History of botulinum toxicity
* Prior scalenectomy
* Surgery for TOS planned within four months
* Use of blood thinners, i.e., warfarin; unfractionated or low molecular weight heparin
* History of Myasthenia Gravis, Eaton-Lambert Syndrome or Shy-Drager Syndrome
* Unable to complete follow-up assessments at 6 weeks and 4 months
* Any abnormalities on EMG, CT or MRI studies suggesting an alternate diagnosis
* Pregnancy or planned pregnancy within six months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Pain | Change from baseline at six weeks and four months
  The primary outcome measure will be change in baseline pain as measured on a ten point Numeric Scale and will be assessed at six weeks and four months following injection.

SECONDARY OUTCOMES:
Paresthesias on Numeric Rating Scale | Change from baseline at six weeks and four months
  Secondary outcomes will be change from baseline in paresthesias as measured on a Numeric Rating Scale at baseline, six weeks and four months.
Function on DASH scale | change from baseline at 6 weeks and 4 monthss
  Secondary outcome will be change from baseline in function on the Disabilities of the arm, shoulder, hand questionnaire at six weeks and at four months.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Finlayson, MD, Principal Investigator — University of British Columbia
Locations (1):
- G F Strong Rehabilitation Centre, Vancouver, British Columbia, Canada